CLINICAL TRIAL: NCT06388226
Title: Leg Heat Therapy to Improve Functional Performance in Heart Failure With Preserved Ejection Fraction (HFpEF)
Brief Title: Leg Heat Therapy in Heart Failure With Preserved Ejection Fraction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Purdue University (Other)
Responsible Party: Principal Investigator, Onyedika Ilonze, Assistant Professor of Clinical Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB # 16143
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Heat therapy (Experimental): Patients will be provided with water-circulating trousers, a water heater, and a water tank coupled to a water pump. The heater will be adjusted to warm up the water to 42ºC. Participants will be asked to apply the therapy daily for 90 min while in the supine position.
  Interventions: Device: Leg heat therapy
- Sham control (Sham Comparator): Patients will be provided with water-circulating trousers, a water heater, and a water tank coupled to a water pump. The heater will be adjusted to warm up the water to 33ºC. Participants will be asked to apply the therapy daily for 90 min while seated or in the supine position.
  Interventions: Device: Leg sham therapy

INTERVENTIONS:
Device: Leg heat therapy — A sous vide heating immersion circulator heats up the water inside the water tank to 42ºC. A water pump circulates temperature-regulated water through the trousers.
  Arms: Heat therapy
Device: Leg sham therapy — A sous vide heating immersion circulator heats up the water inside the water tank to 33ºC. A water pump circulates temperature-regulated water through the trousers.
  Arms: Sham control

SUMMARY:
The objective of this pilot study is to establish evidence to support the validity of HT in improving skeletal muscle function and physical capacity of patients with HFpEF. Our central hypothesis is that HT treatment will lead to improvements in skeletal muscle and microvascular function compared to a control intervention. As a result, we anticipate that patients treated with HT will demonstrate improved skeletal muscle microvascular blood flow and oxygenation resulting in enhanced exercise tolerance. To explore this hypothesis, we propose the following specific aim: Explore the effects of home-based HT on exercise tolerance in patients with HFpEF.

ELIGIBILITY:
Inclusion Criteria:

* Men and women older than 18 years
* Established diagnosis of heart failure with preserved ejection fraction (HFpEF) including left ventricular ejection fraction (LVEF) ≥50% as evidenced by Doppler echocardiography and/or ratio of the early mitral inflow velocity (E) to septal tissue Doppler velocity (e') >8 and at least 1 other sign of chronically elevated filling pressures, including an enlarged left atrium (left atrial volume index >34 mL/m2), an elevated N-terminal pro-brain natriuretic peptide (NT-pro-BNP) level within the past year, long-term loop diuretic use for control of symptoms, or elevated filling pressures (mean pulmonary capillary wedge pressure >12 mmHg) on prior cardiac catheterization
* Stable medical treatment

Exclusion Criteria:

* Recent hospitalization (within the previous 1 month)
* Unstable angina and/or uncontrolled cardiac arrhythmia causing symptoms or hemodynamic compromise (including severe bradycardia or tachycardia, sick sinus syndrome, or multifocal premature ventricular contractions)
* Presence of any clinical condition that makes the patient unsuitable to participate in the trial, e.g., significant ischemic or valvular heart disease, cor pulmonale, unstable coronary artery disease, primary renal (e.g., estimated glomerular filtration rate (eGFR) <25 mL/min/1.73 m2) or hepatic disease (e.g., aspartate aminotransferase and alanine aminotransferase levels >3.0 times the upper limit of the normal range), pulmonary, neuromuscular, orthopedic disorders, among others
* Inability to exercise on the treadmill
* Inability to provide informed consent
* Concern for inability of the patient to comply with study procedures and/or follow up (e.g., alcohol or drug abuse)
* Any contraindication to heat therapy and/or inability to fit into water-circulating trousers
* Impaired thermal sensation in the leg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in time to exhaustion during treadmill exercise | Baseline to 2-month follow-up
  The investigators will determine whether daily leg heat therapy for 90 min using water-circulating trousers perfused with water heated to 42ºC improves the time to exhaustion during treadmill exercise testing at 2-month follow-up compared to a sham treatment.

SECONDARY OUTCOMES:
Change in maximal pulmonary oxygen uptake during treadmill exercise | Baseline to 2-month follow-up
  Maximal pulmonary oxygen uptake (VO2max) will be evaluated during treadmill exercise testing. The investigators will determine whether leg heat therapy improves VO2max at 2-month follow-up compared to the sham treatment.
Change in triceps surae microvascular oxygenation during treadmill exercise | Baseline to 2-month follow-up
  Microvascular oxygenation will be assessed using near-infrared spectroscopy (NIRS) during treadmill exercise testing. The investigators will determine whether leg heat therapy improves muscle microvascular oxygenation at 2-month follow-up compared to the sham treatment.
Change in systolic blood pressure | Baseline to 2-month follow-up
  The systolic blood pressure will be measured in triplicate using a blood pressure monitor. The investigators will determine whether leg heat therapy improves systolic blood pressure at 2-month follow-up compared to the sham treatment.
Change in diastolic blood pressure | Baseline to 2-month follow-up
  The diastolic blood pressure will be measured in triplicate using a blood pressure monitor. The investigators will determine whether leg heat therapy improves blood pressure at 2-month follow-up compared to the sham treatment.
Change in Minnesota Living with Heart Failure Questionnaire (MLHFQ) score | Baseline to 2-month follow-up
  Health-related quality of life will then be assessed via the MLHFQ, which is a validated, self-administered, 21-item disease-specific instrument for patients with heart failure. Items are scored in a 6-point Likert scale (0 to 5) and reflect physical, emotional and socioeconomic status during the past 4 weeks. The questionnaire is scored by summation of all 21 responses (with higher scores indicating poorer quality of life).
Change in triceps surae microvascular oxygenation during reactive hyperemia | Baseline to 2-month follow-up
  Microvascular oxygenation will be assessed using near-infrared spectroscopy (NIRS) during reactive hyperemia. The investigators will determine whether leg heat therapy improves muscle microvascular oxygenation at 2-month follow-up compared to the sham treatment.
Change in triceps surae volume | Baseline to 2-month follow-up
  The volume of calf muscles will be determined using magnetic resonance (MR) images. The investigators will determine whether leg heat therapy improves calf muscle volume at 2-month follow-up compared to the sham treatment.
Change in triceps surae intramuscular fat content | Baseline to 2-month follow-up
  The intramuscular fat content of calf muscles will be determined using magnetic resonance (MR) images. The investigators will determine whether leg heat therapy reduces intramuscular fat content at 2-month follow-up compared to the sham treatment.
Change in the time constant for phosphocreatine recovery after dynamic exercise | Baseline to 2-month follow-up
  Magnetic resonance spectroscopy tuned to phosphorous (31PMRS) will be used to measure the time constant for PCr recovery (τ) after dynamic planar flexion exercise. The investigators will determine whether leg heat therapy reduces the time constant for PCr recovery at 2-month follow-up compared to the sham treatment.
Change in maximal plantar flexor strength | Baseline to 2-month follow-up
  The maximal voluntary contraction (MVC) strength of the plantar flexor muscles will be assessed using an MR-compatible ergometer. Participants will be asked to perform three plantar-flexor MVCs separated by a one-minute rest period. The MVC torque will be considered the highest peak torque value measured over the three trials. The investigators will determine whether leg heat therapy improves maximal plantar flexor strength at 2-month follow-up compared to the sham treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - IU Health Methodist, Indianapolis, Indiana
  - IU Health University Hospital, Indianapolis, Indiana